CLINICAL TRIAL: NCT03051815
Title: Influence of Craniofacial Restriction on Rebound of Obstructive Sleep Apnea Following Weight Gain
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Susanna SS Ng, Honorary Assistant Professor, Chinese University of Hong Kong
Other Study IDs: OSA-MMV/Ng/2016
Record Dates: First submitted 2017-02-03; First posted 2017-02-14 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Observation
Keywords: obstructive sleep apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Apart from obesity, craniofacial factors are well recognized in the pathogenesis of obstructive sleep apnea (OSA) and are likely to play an important role in influencing the response to weight loss. The prevalence of OSA syndrome is as common among the middle-aged Hong Kong Chinese populations as the Caucasians, despite our Chinese patients having much lower body mass index (BMI). From previous work on ethnic comparison, for the same degree of OSA severity, Caucasians were more overweight, whereas Chinese exhibited more craniofacial bony restriction. Cephalometric measurements based on lateral radiograph of the upper airway have shown that a shorter distance between maxillary projection from the cranial base, a smaller posterior airway space, less mandibular protrusion, a narrower space between the hard palate and cranial base, and a more caudally placed hyoid bone predispose to a higher apnea-hypopnea index (AHI). A recent study shown that a shorter mandibular length as measured by lateral cephalometry was associated with a greater fall in AHI after weight loss. Another study using craniofacial computed tomography (CT) scans to evaluate the maxillomandibular bony volume found that craniofacial restriction influenced the relationship between weight loss and OSA improvement. Collectively, these studies suggest that the effect on AHI with weight loss is likely to be more pronounced in those with a smaller craniofacial skeleton. However, the effect of the craniofacial restriction on the degree of rebound in OSA following weight gain after the weight loss intervention is unknown.

The study aims to investigate the change in weight and OSA severity following cessation of a lifestyle modification program (LMP) and examine the relationship between craniofacial restriction and the degree of OSA reoccurrence.

DETAILED DESCRIPTION:
All subjects will be advised to stop using continuous positive airway pressure (CPAP) for at least 7 days as previous study showed that severity of obstructive sleep apnea (OSA) did not increase further after the first week of CPAP withdrawal. Subjects will then be invited to undergo a limited sleep study using "EMBLETTA" portable diagnostic system (MEDCARE, Iceland). The EMBLETTA is a pocket-sized digital recording device. It is a multi-channel transducer, providing an apnea-hypopnea index (AHI) based on recording time. It also detects both respiratory and abdominal efforts through the effort sensor and can differentiate between obstructive and central events. Built-in position sensors are also available to differentiate supine from non-supine events. Respiratory events are scored when desaturations of at least 4% occurred in the absence of moving artefacts and irrespective of co-existing changes in snoring or heart rate. The EMBLETTA operates on battery power, with the internal memory storage of 16 MB, which allows approximately 12 hours of data collection. The EMBLETTA default settings for apneas and hypopneas will be used in this study. An apnea is defined as a decrease in airflow by 80% of baseline for at least 10 seconds. The EMBLETTA default maximum apnea duration is set at 80 seconds. A hypopnea is defined as a decrease in airflow by 50% of baseline for at least 10 seconds. The EMBLETTA default maximum hypopnea duration is set at 100 seconds. The EMBLETTA AHI used for analysis is automatically analysed by the EMBLETTA software. The EMBLETTA device has been validated against hospital-based polysomnography in the Hong Kong Chinese population. The EMBLETTA is a highly sensitive and specific screening device in quantifying AHI and differentiating obstructing and supine events when compared against polysomnography (PSG) in patients with suspected OSA. Patients will be instructed how to operate the EMBLETTA device for the sleep recording and estimate their time of sleep. Those who have failed the EMBLETTA sleep study will be arranged to have a second home EMBLETTA sleep study. Patients who are symptomatic of OSA with a negative home EMBLETTA sleep study will be arranged to have a hospital-based PSG.

All subjects will undergo three-dimensional (3D) computed tomography (CT) scans of the head/neck region to evaluate the upper airway and craniofacial structures. Craniofacial restriction is determined by measuring the size of the maxillomandibular volume based on the mandibular cephalometric landmarks (left and right condylion, left and right gonion, anterior nasal spine (ANS) and menton) as per previous published study. The patient is positioned in the natural head position with a closed lip and bite. All measurements will be made by a single assessor and the analysis will be performed blind to knowledge of weight loss and AHI data.

All subjects will go through several measurements. These include assessment of subjective sleepiness with the Epworth Sleepiness scale (ESS), anthropometric measurements (body mass index, neck and waist circumference) and blood pressure.

The ESS is a questionnaire specific to symptoms of daytime sleepiness and the patients are asked to score the likelihood of falling asleep in eight different situations with different levels of stimulation, adding up to a total score of 0 to 24.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are participants in a previously described dietician-based weight loss study in obese Chinese with obstructive sleep apnea (OSA). Specific study entry criteria included an age range between 30 and 80 years, body mass index (BMI) >25 kg/m2, and moderate to severe OSA (apnea-hypopnea index (AHI) >15 events/hour) before the weight loss program performed in the year of 2010-2013.

Exclusion Criteria:

* Subjects refused to participate the trial or unable to consent.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects are participants in a previously described dietician-based weight loss study in obese Chinese with obstructive sleep apnea (OSA) in which 61 subjects underwent a 12-month weight loss program consisting of dietician consultation with caloric reduction of 10% to 20% in daily energy intake from the patient's usual diet and then the goal was adjusted subsequently based on changes in body weight with target BMI toward 23 kg/m2 om the uear pf 2010-2013. Specific study entry criteria included an age range between 30 and 80 years, body mass index (BMI) >25 kg/m2, and moderate to severe OSA (apnea-hypopnea index (AHI) >15/hr) before the weight loss program performed in the year of 2010-2013. All subjects from the intervention group will be invited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Change in apnea-hypopnea index (AHI) | 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Susanna So-Shan Ng, MBChB, Principal Investigator — Hospital Authority
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No